CLINICAL TRIAL: NCT01718366
Title: Phase I-II Study of Association of Deferasirox, Vitamin D and Azacytidine as Treatment of High Risk MDS (IPSS Int-2 and High)
Brief Title: A Study of Combined Deferasirox, Vitamin D and Azacytidine in High Risk MDS
Acronym: GFM-EXVD-AZA
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Groupe Francophone des Myelodysplasies (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GFM-EXVD-AZA-2011-005623-41
Record Dates: First submitted 2012-10-24; First posted 2012-10-31 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: MDS
MeSH Terms: interventions — Deferasirox; Vitamin D; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ferritin level >300ng/ml and < 1000ng/ml (Experimental): Patients will be included in 2 groups according to the ferritin level at time of inclusion.
  Patients with the ferritin level >300ng/ml and < 1000ng/ml, will be included in Group 1.
  Interventions: Deferasirox, Vitamin D (100000/week) and Azacitidine (75 mg/kg/day Day1 today 7)
  5 patients in each cohort: Cohort 1: Deferasirox: 5mg/kg/d Cohort 2: Deferasirox: 10mg/kg/d Cohort 3: Deferasirox: 15mg/kg/d
  Interventions: Drug: Deferasirox, Vitamin D and Azacitidine
- ferritin level > 1000ng/ml (Experimental): Patients will be included in 2 groups according to the ferritin level at time of inclusion.
  Patients with the ferritin level > 1000ng/ml, will be included in Group 2. Intervention: Deferasirox, Vitamin D (100000/week) and Azacitidine (75 mg/kg/day Day1 today 7)
  5 patients in each cohort: Cohort 1: Deferasirox: 10mg/kg/d Cohort 2: Deferasirox: 15mg/kg/d Cohort 3: Deferasirox: 20mg/kg/d
  Interventions: Drug: Deferasirox, Vitamin D and Azacitidine

INTERVENTIONS:
Drug: Deferasirox, Vitamin D and Azacitidine — association of Deferasirox (group 1: 5-10-15/mg/kg/day according to dose level group), Vitamine D (100000U/week) and Azacitidine (75 mg/kg/day day1-day7)
  Other Names: Exjade; VitaminD; Vidaza

SUMMARY:
Determinate safety and response rate of the association Deferasirox -Vitamine D - Azacitidine in treatment of high risk MDS

Deferasirox Exjade:

The dose of Deferasirox will be assigned according to the ferritin level. Dose escalation is scheduled during the phase I, with 5 additional patients per group.

The maximal tolerated dose of Deferasirox will be required for the phase II of the study.

The first dose will be assigned according to the ferritin level of the patient at time of inclusion:

5 mg/kg/d if the ferritin is >300ng/ml and < 1000ng/ml in Group 1 10 mg/kg/d if the ferritin is ≥1000ng/ml) in Group 2

Group 1 : Ferritin 300 to 1000ng /ml:

* cohort 1 : 5 mg/kg/d
* cohort 2 : 10mg/kg/d
* cohort 3 : 15 mg/kg/d

Group 2 : Ferritin > 1000ng /ml:

* cohort 1 : 10 mg/kg/d
* cohort 2 : 15mg/kg/d
* cohort 3 : 20 mg/kg/d

  5 patients will be treated by cohort. In absence of toxicity (extra-hematological toxicity grade 3 or 4 or hematological grade 4), 5 additional patients will be included in the next cohort.

Deferasirox will be administrated once daily during all the study period. Uvedose will be administrated once weekly during all the study period (100.000 UI P.O).

Azacitidine will be administrated sc at 75 mg/m²/d, during 7 days, J1 to J7 of each cycles(One cycle is 28 days)

During phase I and II, Deferasirox will always be associated with Vitamin D and Azacitidine

Patients will be received 6 cycles of treatment (except if progression, unacceptable toxicity or withdrawn of patients occured) After 3 and 6 cycles, an evaluation will be done to evaluate the efficacy of the treatment.

No dose modification of deferasirox will be done after 3 cycles of treatment except in case of progression). After 6 cycles, patients with CR, PR, marrow CR or HI will be treated with the same dose of Deferasirox until progression .

DETAILED DESCRIPTION:
Deferasirox will be administrated once daily in the morning on an empty stomach, 30 minutes before meal.

Deferasirox will be stopped if the ferritin level is under 100 ng/ml,and could be restarted is the ferritin level increase to 200 ng/ml

Uvedose dose could be adjusted according to the phosphocalcic metabolism parameters and the plasma Vitamin D3 level.

ELIGIBILITY:
Inclusion Criteria:

* High risk MDS, according to OMS classification
* High risk CMML (WBC < 13 G/L)
* AREBT of the FAB classification with less than 30% of blastes
* IPSS>=1.5 (int-2 and high risk)
* Age >=18y
* Performance status<=2 (ECOG)
* Bilirubin and transaminase < 1.5 x ULN
* Normal renal function
* Patient not eligible for Allogeneic stem cell transplant
* Male and female patients must use an effective contraceptive method during the study and for a minimum of 3 months after study treatment.
* Agree the need for the use of a condom if engaged in sexual activity with a pregnant woman or a woman of childbearing potential. during the entire period of treatment, even if disruption of treatment and during 3 months after end of treatment
* Male patient: Agree not to conceive during treatment and study drug therapy (including doses interruptions) and for 3 months after the end of the study drug therapy
* Agree not to donate semen during study drug therapy and for one week after end of study drug therapy.
* Agree to learn about the procedures for preservation of sperm,before starting treatment
* Patient be able to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

* Active infection or uncontrolled disease
* Use of cytotoxic chemotherapeutic agents or experimental agents(agents that are not commercially available) for the treatment of MDS within 28 days. In case of used of cytotoxic chemotherapeutic agents or hypomethylating agent a wash out of 3 mont is required.
* Active Cancer or Cancer within one year before inclusion
* Previous calcic urinary lithiasis
* Previous hyperparathyroid primitive disease or uncontrolled
* Hypercalcemia, hyperphosphoremia, hypervitaminosis D
* Patient already include in another experimental study
* Active infection by HIV, hepatite B or C
* Pregnant or lactating females
* Patient not able (medical/psychiatric) to understand and sign the written consent
* Patients with a ferritin level less than 300ng/ml
* Patient eligible for an Allogeneic stem cell transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
To determine the maximal tolerated dose(MTD | 6 month of treatment
  patient will be evaluable after at least one cycle. Treatment will be administrated during 6 month and responders will be treated until progression or death

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Hermine, MD, Principal Investigator — Necker Hospital (Paris); Pierre Fenaux, MD, Study Director — Saint Louis Hospital (Paris); Felipe Suarez, MD, Study Chair — Necker Hospital (Paris)
Locations (15):
- GENT, Ghent, Belgium
- France (14):
  - Centre Hospitalier de La Cote Basque, Bayonne
  - Hôpital Avicenne, Bobigny
  - Centre Hospitalier de Boulogne sur Mer, Boulogne-sur-Mer
  - CHU Le Mans, Le Mans
  - Hôpital Saint Vincent de Paul, Lille
  - CHU Limoges, Limoges
  - CHU Brabois, Nancy
  - CHU Nantes, Nantes
  - Centre Catherine de Sienne, Nantes
  - Hôpital saint Louis, Paris
  - Hôpital cochin, Paris
  - Hôpital Necker, Paris
  - CHU Poitiers, Poitiers
  - IUCT Oncopole Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No